CLINICAL TRIAL: NCT04348435
Title: A Randomized, Double-Blind, Placebo-Controlled, Clinical Trial to Assess Efficacy and Safety of Allogeneic HB-adMSCs to Provide Immune Support Against COVID-19.
Brief Title: A Randomized, Double-Blind, Single Center, Efficacy and Safety Study of Allogeneic HB-adMSCs Against COVID-19.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HBCOV02
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Results first posted 2022-11-17 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: Coronavirus; Prevention; Immune support; stem cells; mesenchymal stem cells; adipose-derived mesenchymal stem cells
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Allogeneic HB-adMSCs 200MM (Experimental): Subjects assigned to this arm will receive 5 intravenous infusions of HB-adMSCs at 200 million cells/dose. Infusions will occur at weeks 0, 2, 6, 10, and 14.
  Interventions: Biological: HB-adMSCs
- Allogeneic HB-adMSCs 100MM (Experimental): Subjects assigned to this arm will receive 5 intravenous infusions of HB-adMSCs at 100 million cells/dose. Infusions will occur at weeks 0, 2, 6, 10, and 14.
  Interventions: Biological: HB-adMSCs
- Allogeneic HB-adMSCs 50MM (Experimental): Subjects assigned to this arm will receive 5 intravenous infusions of HB-adMSCs at 50 million cells/dose. Infusions will occur at weeks 0, 2, 6, 10, and 14.
  Interventions: Biological: HB-adMSCs
- Placebo (Placebo Comparator): Subjects assigned to this arm will receive 5 intravenous infusions of placebo intervention (saline). Infusions will occur at weeks 0, 2, 6, 10, and 14.
  Interventions: Other: Placebos

INTERVENTIONS:
Biological: HB-adMSCs — Hope Biosciences allogeneic adipose-derived mesenchymal stem cells
  Arms: Allogeneic HB-adMSCs 100MM; Allogeneic HB-adMSCs 200MM; Allogeneic HB-adMSCs 50MM
Other: Placebos — Saline
  Arms: Placebo

SUMMARY:
Hope Biosciences is conducting a research study of an investigational product called allogeneic adipose-derived mesenchymal stem cells (abbreviated as HB-adMSCs) to provide immune support against COVID-19. The study purpose is to evaluate the safety and efficacy of five IV infusions of HB-adMSCs in subjects with no signs of COVID-19.

DETAILED DESCRIPTION:
This is a Phase II, Randomized, Placebo-Controlled, Double-Blinded, Clinical Trial to Assess Efficacy of HB-adMSCs to Provide Immune Support Against Coronavirus Disease. 100 patients will be enrolled. Eligible participants are at high or very high exposure risk of contracting COVID-19. The primary endpoint of this study is to provide immune support against COVID-19, measured by the percentage of subjects that develop symptoms of COVID-19. In addition, participants will be monitored for overall clinical status by standard clinical laboratories and inflammatory markers. Participants will complete Short Form Health Survey (SF-36) and depression module (PHQ-9) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Men, and women 18 years of age or older
* Participant works in a capacity that is characterized as high-risk or very high-risk
* High-Risk Exposure jobs are those with high potential for exposure to known or suspected sources of COVID-19.
* First responders, health care delivery and support staff (e.g., law enforcement, fire fighters, paramedics, doctors, nurses, and other hospital staff who must enter patients' rooms) exposed to individuals potentially having COVID-19.
* Mortuary workers involved in preparing (e.g., for burial or cremation) the bodies of people who are known to have, or suspected of having, COVID-19 at the time of their death
* Very High-Risk Exposure jobs are those with high potential for exposure to known or suspected sources of COVID-19 during specific medical, postmortem or laboratory procedures.
* Health care workers (e.g., doctors, nurses, dentists, paramedics, emergency medical technicians) performing aerosol-generating procedures (e.g., intubation, cough induction procedures, bronchoscopies, some dental procedures and exams or invasive specimen collection) on known or suspected COVID-19 patients.
* Health care or laboratory personnel collecting or handling specimens from known or suspected COVID-19 patients (e.g., manipulating cultures from known or suspected COVID-19 patients).
* Morgue workers performing autopsies, which generally involve aerosol-generating procedures, on the bodies of people who are known to have, or suspected of having, COVID-19 at the time of their death
* No signs or symptoms of infection, including but not limited to, body temperature >100 F and pulse rate > 100 BPM.
* Subject provides written informed consent prior to initiation of any study procedures.--Agrees to the collection of venous blood per protocol.
* Agrees to conformational testing for SARS-CoV-2 before end of study.

Exclusion Criteria:

* Women who are pregnant or lactating, or those who are not pregnant but do not take effective contraceptive measures
* Patients who are participating in other clinical trials or have intake of investigational drug within the previous 30 days;
* Inability to provide informed consent or to comply with test requirements;
* Any medical disease or condition that, in the opinion of the site PI or sub-investigator, precludes study participation. Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
* Patients who have received a stem cell treatment within one year.
* Receipt of any other SARS-CoV-2 or other experimental coronavirus vaccine at any time prior to or during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Cheng, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Selection of subjects was based on the inclusion and exclusion criteria and only those subjects who met all of the inclusion criteria and none of the exclusion criteria, were eligible to participate in the trial. The first participant was enrolled on 05/14/2020 and the last participant was enrolled on 11/04/2020.
Pre-assignment Details: A total of 84 subjects were assessed for screening, out of which only 53 were enrolled and 31 were screen failed.
Groups:
- Allogeneic HB-adMSCs 200MM: Subjects assigned to this arm will receive 5 intravenous infusions of HB-adMSCs at 200 million cells/dose.
  HB-adMSCs: Hope Biosciences allogeneic adipose-derived mesenchymal stem cells
- Allogeneic HB-adMSCs 100MM: Subjects assigned to this arm will receive 5 intravenous infusions of HB-adMSCs at 100 million cells/dose.
  HB-adMSCs: Hope Biosciences allogeneic adipose-derived mesenchymal stem cells
- Allogeneic HB-adMSCs 50MM: Subjects assigned to this arm will receive 5 intravenous infusions of HB-adMSCs at 50 million cells/dose.
  HB-adMSCs: Hope Biosciences allogeneic adipose-derived mesenchymal stem cells
- Placebo: Subjects assigned to this arm will receive 5 intravenous infusions of placebo intervention (saline).
  Placebos: Saline
Period: Overall Study
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
Started | 19 | 9 | 12 | 13
Completed | 11 | 5 | 9 | 10
Not Completed | 8 | 4 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo | Total
Number analyzed (Participants) | 19 | 9 | 12 | 13 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (13.34) | 47.6 (9.65) | 43.9 (12.38) | 42.8 (9.97) | 44.9 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 7 | 8 | 30
  Male | 9 | 4 | 5 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 4 | 11
  Not Hispanic or Latino | 16 | 7 | 10 | 9 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 2 | 1 | 7
  White | 13 | 8 | 7 | 10 | 38
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 9 | 12 | 13 | 53
Height [Mean (Standard Deviation); unit: cm] | 172.05 (10.18) | 167.35 (11.60) | 168.38 (8.70) | 171.54 (11.66) | 170.30 (10.39)
Body Weight [Mean (Standard Deviation); unit: kg] | 93.132 (29.12) | 85.982 (26.72) | 78.662 (14.69) | 79.763 (23.51) | 85.362 (24.84)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.14 (8.426) | 30.18 (6.271) | 27.61 (3.946) | 26.83 (6.606) | 29.12 (6.893)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Were Hospitalized Due to COVID-19 Symptoms
Description: Number of subjects that were hospitalized due to COVID-19 symptoms during the conduct of this study.
Time Frame: Week 0 through Week 26 (End of Study)
Population: A total of 37 subjects completed all 5 infusions.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
Number analyzed (Participants) | 13 | 5 | 10 | 9
Participants
  Number of Subjects that were Hospitalized due to COVID-19 Symptoms | 0 | 0 | 0 | 0
  Number of Subjects that were not Hospitalized due to COVID-19 Symptoms | 13 | 5 | 10 | 9

2. Primary Outcome: Number of Participants That Had Symptoms Associated With COVID-19
Description: Number of subjects who experience symptoms defined to be associated with COVID-19, such as fever, shortness of breath/difficulty breathing, cough, etc.
Time Frame: Week 0 through Week 26 (End of Study)
Population: A total of 37 subjects who completed all 5 infusions.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
Number analyzed (Participants) | 13 | 5 | 10 | 9
Participants
  Number of Subjects with Incidence of COVID-19 Symptoms | 4 | 0 | 0 | 0
  Number of Subjects with No Incidence of COVID-19 Symptoms | 9 | 5 | 10 | 9

3. Secondary Outcome: Leukocyte Differential Count
Description: Change from baseline in Leukocyte Differential Count
Time Frame: Week 0 to Week 26 (End of Study)
Population: Number of subjects contributing to analysis.
Measure: Least Squares Mean (Standard Error); unit: Leukocytes (x10^9/L)
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
Number analyzed (Participants) | 11 | 4 | 6 | 6
Leukocytes (x10^9/L)
  LSMeans | 6.204 (0.296) | 5.518 (0.502) | 6.029 (0.393) | 5.951 (0.392)
  Change from baseline | 0.508 (0.296) | -0.179 (0.502) | 0.333 (0.393) | 0.255 (0.392)
Statistical Analysis 1: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Test type: Superiority; p = 0.6113, ANCOVA; Mean Difference (Net) = 0.253, Standard Error of Mean 0.490
Statistical Analysis 2: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Test type: Superiority; p = 0.5039, ANCOVA; Mean Difference (Net) = -0.434, Standard Error of Mean 0.638
Statistical Analysis 3: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Test type: Superiority; p = 0.8903, ANCOVA; Mean Difference (Net) = 0.077, Standard Error of Mean 0.555

4. Secondary Outcome: C Reactive Protein
Description: Change from baseline in C Reactive Protein
Time Frame: Week 0 through Week 26 (End of Study)
Population: Number of subjects contributing to analysis.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
Number analyzed (Participants) | 11 | 4 | 6 | 6
mg/L
  LSMeans | 2.424 (0.632) | 1.759 (1.047) | 2.679 (0.846) | 2.671 (0.843)
  Change from baseline | -0.609 (0.632) | -1.275 (1.047) | -0.354 (0.846) | -0.362 (0.843)
Statistical Analysis 1: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Test type: Superiority; p = 0.8171, ANCOVA; Mean Difference (Net) = -0.247, Standard Error of Mean 1.056
Statistical Analysis 2: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Test type: Superiority; p = 0.5034, ANCOVA; Mean Difference (Net) = -0.913, Standard Error of Mean 1.342
Statistical Analysis 3: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Test type: Superiority; p = 0.9948, ANCOVA; Mean Difference (Net) = 0.008, Standard Error of Mean 1.193

5. Secondary Outcome: Tumor Necrosis Factor - Alpha
Description: Change from baseline in TNF alpha
Time Frame: Week 0 through Week 26 (End of Study)
Population: Number of subjects contributing to analysis.
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
Number analyzed (Participants) | 11 | 4 | 6 | 6
ng/L
  LSMeans | 1.175 (0.091) | 0.951 (0.150) | 1.173 (0.123) | 0.996 (0.124)
  Change from baseline | -0.316 (0.091) | -0.540 (0.150) | -0.318 (0.123) | -0.495 (0.124)
Statistical Analysis 1: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Test type: Superiority; p = 0.2641, ANCOVA; Mean Difference (Net) = 0.179, Standard Error of Mean 0.156
Statistical Analysis 2: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Test type: Superiority; p = 0.8220, ANCOVA; Mean Difference (Net) = -0.045, Standard Error of Mean 0.198
Statistical Analysis 3: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Test type: Superiority; p = 0.3097, ANCOVA; Median Difference (Net) = 0.178, Standard Error of Mean 0.171

6. Secondary Outcome: Interleukin 6
Description: Change from baseline in IL-6
Time Frame: Week 0 through Week 26 (End of Study)
Population: Number of subjects contributing to analysis.
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
Number analyzed (Participants) | 11 | 4 | 6 | 6
ng/L
  LSMeans | 1.620 (0.040) | 1.620 (0.065) | 1.732 (0.053) | 1.620 (0.056)
  Change from baseline | -0.019 (0.040) | -0.019 (0.065) | 0.092 (0.053) | -0.019 (0.056)
Statistical Analysis 1: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Test type: Superiority; p = 1.000, ANCOVA; Mean Difference (Net) = 0.000, Standard Error of Mean 0.070
Statistical Analysis 2: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Test type: Superiority; p = 1.000, ANCOVA; Mean Difference (Net) = 0.000, Standard Error of Mean 0.087
Statistical Analysis 3: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Test type: Superiority; p = 0.1713, ANCOVA; Mean Difference (Net) = 0.112, Standard Error of Mean 0.079

7. Secondary Outcome: Interleukin 10
Description: Change from baseline in IL-10
Time Frame: Week 0 through Week 26 (End of Study)
Population: Number of subjects contributing to analysis.
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
Number analyzed (Participants) | 11 | 4 | 6 | 6
ng/L
  LSMeans | 0.768 (0.054) | 0.680 (0.089) | 0.680 (0.073) | 0.688 (0.073)
  Change from baseline | 0.088 (0.054) | 0.000 (0.089) | 0.000 (0.073) | 0.008 (0.073)
Statistical Analysis 1: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Test type: Superiority; p = 0.3868, ANCOVA; Mean Difference (Net) = 0.080, Standard Error of Mean 0.091
Statistical Analysis 2: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Test type: Superiority; p = 0.9429, ANCOVA; Mean Difference (Net) = -0.008, Standard Error of Mean 0.115
Statistical Analysis 3: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Test type: Superiority; p = 0.9362, ANCOVA; Mean Difference (Net) = -0.008, Standard Error of Mean 0.103

8. Secondary Outcome: Short Form-36 (SF-36)
Description: The Short Form-36 Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores (including Energy/Fatigue scores, Social Functioning, role limitations due to Physical Health, General Health, Physical Functioning, Pain, Emotional Well-Being, and Emotional Problems) which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Time Frame: Week 0 to Week 26 (End of Study)
Population: Number of subjects contributing to analysis.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
Number analyzed (Participants) | 11 | 4 | 9 | 8
Score on a Scale
  Average Energy/Fatigue | 68.858 (5.139) | 78.346 (7.672) | 75.849 (5.125) | 69.567 (5.826)
  Average Energy/Fatigue - Change from baseline | 7.140 (5.139) | 16.628 (7.672) | 14.130 (5.125) | 7.848 (5.826)
  Average Social Functioning | 98.950 (2.190) | 90.711 (3.556) | 99.864 (2.503) | 98.430 (2.484)
  Average Social Functioning - Change from baseline | 7.153 (2.190) | -1.086 (3.556) | 8.067 (2.503) | 6.633 (2.484)
  Avg. Role Limitations Due to Physical Health | 94.711 (2.326) | 100.00 (4.393) | 98.727 (2.587) | 98.831 (2.737)
  Avg. Role Limitations Due to Physical Health - Change from baseline | 1.742 (2.326) | 14.280 (4.393) | 5.758 (2.587) | 5.862 (2.737)
  Average General Health | 76.481 (3.818) | 78.857 (6.274) | 81.016 (4.196) | 75.518 (4.454)
  Average General Health - Change from baseline | 1.481 (3.818) | 3.857 (6.274) | 6.016 (4.196) | 0.518 (4.454)
  Average Physical Functioning | 92.361 (2.660) | 96.806 (4.420) | 93.598 (2.939) | 89.928 (3.123)
  Average Physical Functioning - Change from baseline | 1.267 (2.660) | 5.712 (4.420) | 2.504 (2.939) | -1.166 (3.123)
  Average Pain | 90.744 (3.746) | 84.700 (6.291) | 91.166 (4.124) | 79.065 (4.377)
  Average Pain - Change from baseline | 11.212 (3.746) | 5.169 (6.291) | 11.635 (4.124) | -0.466 (4.377)
  Average Emotional Well Being | 87.057 (2.566) | 88.413 (4.096) | 86.992 (2.739) | 84.724 (2.863)
  Average Emotional Well Being - Change from baseline | 4.057 (2.566) | 5.413 (4.096) | 3.992 (2.739) | 1.724 (2.863)
  Avg. Role Limitations Due to Emotional Problems | 99.667 (2.334) | 97.000 (3.654) | 97.000 (2.456) | 97.000 (2.601)
  Avg. Role Limitations Due to Emotional Problems - Change from baseline | 3.833 (2.334) | 1.166 (3.654) | 1.166 (2.456) | 1.166 (2.601)
Statistical Analysis 1: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Average Energy/Fatigue - Treatment Contrast; Test type: Superiority; p = 0.9333, ANCOVA; Mean Difference (Net) = -0.708, Standard Error of Mean 8.380
Statistical Analysis 2: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Average Energy/Fatigue - Treatment Contrast; Test type: Superiority; p = 0.3627, ANCOVA; Mean Difference (Net) = 8.780, Standard Error of Mean 9.483
Statistical Analysis 3: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Average Energy/Fatigue - Treatment Contrast; Test type: Superiority; p = 0.4160, ANCOVA; Mean Difference (Net) = 6.282, Standard Error of Mean 7.604
Statistical Analysis 4: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Average Social Functioning - Treatment Contrast; Test type: Superiority; p = 0.8768, ANCOVA; Mean Difference (Net) = 0.520, Standard Error of Mean 3.320
Statistical Analysis 5: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Average Social Functioning - Treatment Contrast; Test type: Superiority; p = 0.0869, ANCOVA; Mean Difference (Net) = -7.719, Standard Error of Mean 4.344
Statistical Analysis 6: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Average Social Functioning - Treatment Contrast; Test type: Superiority; p = 0.6864, ANCOVA; Mean Difference (Net) = 1.434, Standard Error of Mean 3.514
Statistical Analysis 7: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Avg. Role Limitations Due to Physical Health - Treatment Contrast; Test type: Superiority; p = 0.2587, ANCOVA; Mean Difference (Net) = -4.120, Standard Error of Mean 3.571
Statistical Analysis 8: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Avg. Role Limitations Due to Physical Health - Treatment Contrast; Test type: Superiority; p = 0.1250, ANCOVA; Mean Difference (Net) = 8.417, Standard Error of Mean 5.316
Statistical Analysis 9: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Avg. Role Limitations Due to Physical Health - Treatment Contrast; Test type: Superiority; p = 0.9780, ANCOVA; Mean Difference (Net) = -0.104, Standard Error of Mean 3.732
Statistical Analysis 10: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Average General Health - Treatment Contrast; Test type: Superiority; p = 0.8721, ANCOVA; Mean Difference (Net) = 0.963, Standard Error of Mean 5.925
Statistical Analysis 11: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Average General Health - Treatment Contrast; Test type: Superiority; p = 0.6694, ANCOVA; Mean Difference (Net) = 3.340, Standard Error of Mean 7.735
Statistical Analysis 12: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Average General Health - Treatment Contrast; Test type: Superiority; p = 0.3733, ANCOVA; Mean Difference (Net) = 5.498, Standard Error of Mean 6.073
Statistical Analysis 13: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Average Physical Functioning - Treatment Contrast; Test type: Superiority; p = 0.5594, ANCOVA; Mean Difference (Net) = 2.433, Standard Error of Mean 4.116
Statistical Analysis 14: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Average Physical Functioning - Treatment Contrast; Test type: Superiority; p = 0.2127, ANCOVA; Mean Difference (Net) = 6.878, Standard Error of Mean 5.389
Statistical Analysis 15: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Average Physical Functioning - Treatment Contrast; Test type: Superiority; p = 0.4012, ANCOVA; Mean Difference (Net) = 3.670, Standard Error of Mean 4.303
Statistical Analysis 16: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Average Pain - Treatment Contrast; Test type: Superiority; p = 0.0521, ANCOVA; Mean Difference (Net) = 11.678, Standard Error of Mean 5.748
Statistical Analysis 17: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Average Pain - Treatment Contrast; Test type: Superiority; p = 0.4704, ANCOVA; Mean Difference (Net) = 5.635, Standard Error of Mean 7.696
Statistical Analysis 18: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Average Pain - Treatment Contrast; Test type: Superiority; p = 0.0544, ANCOVA; Mean Difference (Net) = 12.101, Standard Error of Mean 6.017
Statistical Analysis 19: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Average Emotional Well Being - Treatment Contrast; Test type: Superiority; p = 0.5535, ANCOVA; Mean Difference (Net) = 2.333, Standard Error of Mean 3.888
Statistical Analysis 20: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Average Emotional Well Being - Treatment Contrast; Test type: Superiority; p = 0.4642, ANCOVA; Mean Difference (Net) = 3.689, Standard Error of Mean 4.969
Statistical Analysis 21: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Average Emotional Well Being - Treatment Contrast; Test type: Superiority; p = 0.5692, ANCOVA; Mean Difference (Net) = 2.268, Standard Error of Mean 3.936
Statistical Analysis 22: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Avg. Role Limitations Due to Emotional Problems - Treatment Contrast; Test type: Superiority; p = 0.4642, ANCOVA; Median Difference (Net) = 2.667, Standard Error of Mean 3.592
Statistical Analysis 23: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Avg. Role Limitations Due to Emotional Problems - Treatment Contrast; Test type: Superiority; p = 1.0000, ANCOVA; Mean Difference (Net) = 0.000, Standard Error of Mean 4.444
Statistical Analysis 24: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Avg. Role Limitations Due to Emotional Problems - Treatment Contrast; Test type: Superiority; p = 1.0000, ANCOVA; Mean Difference (Net) = 0.000, Standard Error of Mean 3.526

9. Secondary Outcome: Patient Health Questionnaire (PHQ-9) Scores
Description: The study used PHQ-9 as a depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day) to monitor the severity of depression.
Time Frame: Week 0 to Week 26 (End of Study)
Population: Number of subjects contributing to analysis.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
Number analyzed (Participants) | 11 | 3 | 9 | 8
Score on a Scale
  LSMeans | 1.373 (0.489) | 0.912 (0.763) | 1.114 (0.456) | 1.517 (0.538)
  Change from baseline | -1.111 (0.489) | -1.572 (0.763) | -1.370 (0.456) | -0.967 (0.538)
Statistical Analysis 1: Comparison: Allogeneic HB-adMSCs 200MM vs Placebo; Test type: Superiority; p = 0.8628, ANCOVA; Mean Difference (Net) = -0.144, Standard Error of Mean 0.825
Statistical Analysis 2: Comparison: Allogeneic HB-adMSCs 100MM vs Placebo; Test type: Superiority; p = 0.5257, ANCOVA; Mean Difference (Net) = -0.605, Standard Error of Mean 0.940
Statistical Analysis 3: Comparison: Allogeneic HB-adMSCs 50MM vs Placebo; Test type: Superiority; p = 0.5467, ANCOVA; Mean Difference (Net) = -0.403, Standard Error of Mean 0.659

ADVERSE EVENTS:
Time Frame: Week 0 through Week 26 (End of Study)
Description: Out of 53 total subjects, 37 subjects had reported at least one adverse event (AE). A total of 139 AEs were recorded during the entire course of study, out of which 135 were mild in severity, 4 were moderate and none was severe. There were no serious adverse events (SAEs) reported during the study period.
Arm/Group | Allogeneic HB-adMSCs 200MM | Allogeneic HB-adMSCs 100MM | Allogeneic HB-adMSCs 50MM | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/9 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/9 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 15/19 | 5/9 | 7/12 | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic HB-adMSCs 200MM (N=19) | Allogeneic HB-adMSCs 100MM (N=9) | Allogeneic HB-adMSCs 50MM (N=12) | Placebo (N=13)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 2 (2) | 7 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (14) | 2 (3) | 3 (4) | 4 (6)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Influenza like illness (General disorders) | 9 (16) | 2 (4) | 0 (0) | 5 (10)
Fatigue (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary hyper-secretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corona virus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT04348435/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT04348435/SAP_001.pdf